CLINICAL TRIAL: NCT00139152
Title: Exhaled Breath Condensate and Nitric Oxide: Non-invasive Evaluation of Lung Disease After Treatment With Xolair
Brief Title: Non-invasive Ways to Evaluate Lung Disease After Treatment With Xolair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xolair ENO EBC Study
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Lung Disease
Keywords: moderate to severe allergic asthma
MeSH Terms: conditions — Lung Diseases | interventions — Saline Solution; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Placebo
- Xolair (Experimental): Xolair treatment
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Placebo — Saline, Sub-Cuteanous (SQ)
  Other Names: Normal Saline
  Arms: Placebo
Drug: Xolair — Xolair, 0.016 mg/kg Immunoglobulions E (IgE) , SQ
  Other Names: omalizumab; rhumabE25
  Arms: Xolair

SUMMARY:
The purpose of this study is to study the effects of Xolair using non-invasive techniques from the expired gas of patients with moderate to severe allergic asthma.

DETAILED DESCRIPTION:
Traditional methods of sampling secretions from the lower respiratory tract include sputum collection, sputum induction, and bronchoscopy with bronchoalveolar lavage. They cannot be repeated within a short period of time because of their invasiveness, and because the procedures themselves may include an inflammatory response. The need to monitor inflammation in the lungs has led to the exploration of exhaled gases and condensates. Noninvasive monitoring may assist in differential diagnosis of pulmonary diseases, assessment of disease severity and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* On medium to high dose inhaled corticosteroids either with or without a long acting beta agonist
* Baseline IgE 30-700 IU/mL
* Exhaled nitric oxide greater than 13 ppb
* Positive skin test to at least one of the following perennial allergens: cat, dog, dust mite, cockroach
* Stable asthma at the time of enrollment

Exclusion Criteria:

* Concurrent diseases/conditions, history of other diseases/conditions, with clinically significant uncontrolled systemic disease or a history of such disease (eg, infection, hematological, renal, hepatic, coronary heart disease or other cardiovascular disease, endocrinological, or gastrointestinal disease) within previous 3 months
* Upper or lower respiratory tract infection within 6 weeks of screening visit
* Elevated IgE level other than atopy
* Known sensitivity to Xolair
* < 3 months of stable immunotherapy
* Smokers
* Pregnant/nursing women
* Women of childbearing potential who are not practicing medically approved contraceptive methods (eg, oral, subcutaneous, mechanical, or surgical contraception) including abstinence
* Patients who currently hav diagnosed cancer, are currently being investigated for possible cancer or who have any history of cancer
* Known sensitivity to study drug or class of study drugs
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of Xolair on exhaled nitric oxide and leukotriene levels obtained from exhaled breath condensate in patients before and after four months of Xolair or placebo treatment. | post dose

SECONDARY OUTCOMES:
To measure the levels of power of hydrogen (pH), nitrate/nitrite in exhaled breath condensate before and after four months treatment with Xolair and to compare these data to those obtained from the placebo asthmatic control group. | post dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Townley, MD, Principal Investigator — Creighton University Division of Allergy & Immunology; Muhammad A Pasha, M.D., Principal Investigator — Albany Medical CollegeDivision of Allergy, Asthma, & Immunology
Locations (2):
- United States (2):
  - Creighton University Division of Allergy & Immunology, Omaha, Nebraska
  - Albany Medical College, Albany, New York